CLINICAL TRIAL: NCT06527430
Title: Different Local Anesthetic Volumes for Unilateral Spinal Anesthesia in Varicose Vein Surgery
Brief Title: Different Local Anesthetic Volumes for Unilateral Spinal Anesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara Etlik City Hospital (Other Government)
Responsible Party: Principal Investigator, Atakan Sezgi, Principal İnvestigator, Ankara Etlik City Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AEŞH-EK1-2024-0074
Record Dates: First submitted 2024-07-25; First posted 2024-07-30 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-06

CONDITIONS: Discharge Time; Ambulatory Surgery; Spinal Anesthesia
Keywords: local anesthetic volume; varicose vein surgery; ambulatory surgery; spinal anesthesia
MeSH Terms: interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Spinal anesthesia with 4 mg bupivacaine (Active Comparator): After the patients are monitored, they will be placed in the lateral decubitus position. After appropriate field sterilization, patients will undergo unilateral spinal anesthesia with 4 mg bupivacaine. At the fifth minute after spinal anesthesia, patients will be placed in the supine position.
  Interventions: Procedure: 4 mg bupivacaine
- Spinal anesthesia with 6 mg bupivacaine (Active Comparator): After the patients are monitored, they will be placed in the lateral decubitus position. After appropriate field sterilization, patients will undergo unilateral spinal anesthesia with 6 mg bupivacaine. At the fifth minute after spinal anesthesia, patients will be placed in the supine position.
  Interventions: Procedure: 6 mg bupivacaine

INTERVENTIONS:
Procedure: 4 mg bupivacaine — Spinal anesthesia was applied to the patients with 4 mg bupivacaine in the lateral decubitus position.
  Arms: Spinal anesthesia with 4 mg bupivacaine
Procedure: 6 mg bupivacaine — Spinal anesthesia was applied to the patients with 6 mg bupivacaine in the lateral decubitus position.
  Arms: Spinal anesthesia with 6 mg bupivacaine

SUMMARY:
Varicose veins are irreversible and abnormal enlargement of the veins. These veins appear and there are curled swellings under the skin in the feet and legs. Complaints increase when standing and sitting for long periods. For varicose veins in the initial stages, medical treatment methods such as compression socks (elastic socks) and elevating the feet as much as possible can be tried. For widespread varicose veins in more advanced stages, invasive procedures such as sclerotherapy and endovascular ablation are performed. These procedures can be performed under local, spinal or general anesthesia.

Spinal anesthesia; It is a type of neuraxial type of regional anesthesia characterized by injecting local anesthetic drugs into the subarachnoid space alone or together with other drugs, resulting in temporary sensory block, motor block, and sympathetic block. The local anesthetic volume administered during spinal anesthesia may affect the anesthesia levels and discharge times of the patients. For varicose vein surgeries, low-dose local anesthetic is sufficient for spinal anesthesia and can also provide early discharge.

This study will compare the peri-operative effects of different doses of spinal anesthesia in patients undergoing varicose vein surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-80 years
* American Society of Anesthesiologists (ASA) score I-II
* Body Mass Index (BMI) between 18-30 kg/m2
* Patients who underwent spinal anesthesia (bupivacaine 4 mg or 6 mg) for varicose vein surgery in the operating theatre

Exclusion Criteria:

* Patients under 18 and over 80 years of age
* ASA score III and above
* Patients with a history of bleeding diathesis
* Patients with infection in the area to be treated
* BMI below 18 or above 30 kg/m2

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2024-07-30 (Actual); Primary Completion 2025-05-10 (Actual); Study Completion 2025-05-30 (Actual)

PRIMARY OUTCOMES:
Discharge time | On the operation day
  The time (minutes) from the application of spinal anesthesia to the patients' discharge will be recorded as the discharge period.

SECONDARY OUTCOMES:
Motor block appearing time | On the operation day
  Time (minutes) to complete motor block in the lower extremity after spinal anesthesia
Sensorial block appearing time | On the operation day
  Time (minutes) to complete sensorial block in the lower extremity after spinal anesthesia
Motor block disappearing time | On the operation day
  Time (minutes) to disappearance of complete motor block in the lower extremity after spinal anesthesia
Sensorial block disappearing time | On the operation day
  Time (minutes) to disappearance of sensorial block in the lower extremity after spinal anesthesia

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Etlik City Hospital, Yenimahalle, Ankara, Turkey (Türkiye)